CLINICAL TRIAL: NCT05145595
Title: The Effect of Puberty on Pain Sensitivity
Brief Title: Pain Sensitivity During Puberty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Hadas Nahman-Averbuch, Asst Prof of Anesthesiology, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202109120
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Pain
Keywords: Pain; Puberty
MeSH Terms: conditions — Pain | interventions — carboxypeptidase M; Efficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psychophysical assessments of experimental pain (Experimental): At baseline, participants will complete a 2.5-hours study session. In the study session, psychophysical assessments of thermal and pressure stimuli will be performed and sex hormone levels will be analyzed. In addition, demographic, social, pubertal maturation, behavioral and psychological factors will be collected via questionnaires.
  In the optional follow-up portion, participants can complete short surveys every 3 months and/or return for study visits after 6 months and/or after every year depending on the participant's availability. The study visits will include the same procedures as the baseline study visit. Additional surveys regarding new symptoms of pain will be completed. In some cases, participants will meet a pediatric physician who will determine if they meet the criteria for any pain syndrome (for research purposes only).
  Interventions: Device: Thermal Sensory Analyzer; Device: Pressure Stimuli; Device: Mechanical Stimuli; Behavioral: Pain Ratings; Behavioral: Thermal pain thresholds; Behavioral: Pressure pain thresholds (PPT); Behavioral: Mechanical temporal summation; Behavioral: Conditioned pain modulation (CPM) efficiency; Behavioral: Offset analgesia efficiency; Behavioral: Cold pain tolerance

INTERVENTIONS:
Device: Thermal Sensory Analyzer — Thermal stimuli: The Thermal Sensory Analyzer (TSA-II or PATHWAY platform - Medoc, Ramat Yishai, Israel) will be used to deliver heat and cold stimuli. These devices can deliver relatively complex stimuli via computer control. All targeted stimulus temperatures will be less than 50°C, and participants will be free to remove their arm or leg at any time from the thermode. Noxious cold stimuli will also be delivered with a plastic water container or a water bath (FISHER, USA). Participants will be free to pull out of the water bath at any time.
Device: Pressure Stimuli — Pressure stimuli: Pressure stimuli will be applied by using a handheld algometer (Wagner Instruments) or the Pressure Algometer (Medoc, Ramat Yishai, Israel). These devices have a round probe that allows quantifying the amount of pressure that is being applied. The Pressure Algometer allows a real-time visual feedback to control and monitor applied pressure rates. Pressure will be applied to the lower leg, volar forearm, or trapezius.
Device: Mechanical Stimuli — Mechanical stimuli: A set of standardised von Frey filaments (0.25, 0.5, 1, 2, 4, 8, 16, 32, 64, 128 and 256mN). The contact area of the hairs with the skin is of uniform size (<1 mm²) and texture.
Behavioral: Pain Ratings — Pain intensity and pain unpleasantness ratings will be assessed by numerical rating scale (ranging from 0- no pain/unpleasantness to- 100 the most intense/unpleasantness pain imaginable) and by mechanical and computerized visual analog scales (VAS which ranges between ''no pain sensation'' and ''most intense pain imaginable'').
Behavioral: Thermal pain thresholds — Cold and heat pain thresholds (CPT and HPT, respectively) will be determined [22; 55]. Thresholds are determined by continuous ramping of temperature from 32°C baseline temperature until the participant press a button at the first moment he/she feels pain from the stimulus. Cut-off temperatures are 0°C and 50°C, to minimize potential damage to the skin. The baseline temperature to which the thermode returns before each test is 32°C. The first threshold measurement will be used as a familiarization. The average threshold is calculated from three measurements.
Behavioral: Pressure pain thresholds (PPT) — Pressure will be increased continually and participants will be instructed to press a button the first moment they feel pain from the pressure stimulus. The first threshold measurement will be used as a familiarization. The average threshold is calculated from three measurements.
Behavioral: Mechanical temporal summation — A pinprick stimulus with standardised intensity (#6.10 or #6.45 von Frey filament) and a flat contact area of 0.25mm diameter will be used. In this test, participants will rate the pain evoked by a single pinprick stimulus and by a series of 10 identical pinprick stimuli. The 10 identical pinprick stimuli are applied with a frequency of 1 s-1 within an area of 1 cm2. Immediately following the single stimulus and series of stimuli, an evaluation of the pain will be collected. The difference in pain ratings evoked with the one stimuli vs. the 10 stimuli is the temporal summation value.
Behavioral: Conditioned pain modulation (CPM) efficiency — The CPM paradigm assesses endogenous inhibitory pain modulation efficiency related to spatial filtering of nociceptive information. CPM testing includes the application of a "test" stimulus without conditioning (control run) and a subsequent application of the same test stimulus together with a conditioning stimulus (conditioning run). Heat-CPM and pressure-CPM. Heat and pressure CPM will be tested in random order.
  The difference between the pain ratings/thresholds of the test stimulus with vs. without the concomitant conditioning stimulus is the CPM magnitude. CPM<0 (reduction in pain) implies efficient inhibitory pain modulation of spatial filtering.
Behavioral: Offset analgesia efficiency — Offset analgesia (OA) paradigm assesses endogenous inhibitory pain modulation efficiency of temporal filtering of nociceptive information. The mechanisms underlying OA are distinct from the CPM mechanisms [41]. OA is characterized by a disproportionately large reduction in pain perception after a small decrease in temperature during noxious thermal stimulation.
  Offset analgesia will be assessed using the three-temperature method (T1°C 5s, T1+1°C 5s, T1°C 20s). The T1 will be noxious heat (44-48°C) delivered to the hand or leg. During the OA paradigm, real time pain intensity ratings will be obtained using the computerized VAS.
  The difference between the pain ratings of the 10-20 seconds noxious stimulus in the OA paradigm compared to a control paradigm (30 seconds of T1) is the OA magnitude. OA<0 (reduction in pain) implies efficient inhibitory pain modulation of temporal filtering.
Behavioral: Cold pain tolerance — Cold pain tolerance will be assessed by having participants immerse their hand or foot in a cold (4-12°C) water bath. Tolerance will be defined by the time of hand withdrawal. VAS ratings of cold pain intensity might be obtained periodically, and both pain intensity and pain unpleasantness will be recorded upon hand withdrawal. Limb immersion in the cold water bath will be terminated after 120 s if participants do not withdraw their hand before then.

SUMMARY:
Aim 1- To examine the differences in pain sensitivity between adolescents at early vs. mid pubertal status Aim 2- To determine the relationships between sex hormone levels and pain sensitivity Exploratory Aim 1- To determine the effect of pubertal maturation on pain sensitivity Exploratory Aim 2- To identify parameters related to who will develop chronic pain during puberty

Hypothesis 1- Adolescents in early pubertal status will have higher pain ratings and lower pain modulation capabilities compared to adolescents in mid puberal status.

Hypothesis 2- Pain sensitivity will be associated with sex hormone levels. Exploratory Hypothesis 1- As adolescents mature, they will have a decrease in pain sensitivity to experimental pain which will be related to changes in sex hormone levels.

Exploratory hypothesis 2- Female adolescents with greater pain sensitivity, lower testosterone levels and with a family history of pain would be at a higher risk to develop chronic pain

DETAILED DESCRIPTION:
At baseline, participants will complete a 2.5-hours study session. In the study session, psychophysical assessments of thermal and pressure stimuli will be performed and sex hormone levels will be analyzed. In addition, demographic, social, pubertal maturation, behavioral and psychological factors will be collected via questionnaires.

In the optional follow-up portion, participants can complete short surveys every 3 months and/or return for study visits after 6 months and/or after every year depending on the participant's availability. The study visits will include the same procedures as the baseline study visit. Additional surveys regarding new symptoms of pain will be completed. In some cases, participants will meet a pediatric physician who will determine if they meet the criteria for any pain syndrome (for research purposes only).

ELIGIBILITY:
Inclusion Criteria

1. Healthy males and females
2. 9-16 years old
3. English speakers

Exclusion Criteria

Participants will not be enrolled if any of the following criteria exist and based on the investigator discretion:

1. Pregnancy
2. Chronic Pain or frequent headaches (>5 headache /month)
3. Psychiatric or neurological disorders
4. Lack of sensation in the testable limb
5. Disorders associated with pubertal maturation or usage of contraceptive pills that affect sex hormone levels
6. Regular use of pain medications (e.g., opioids, antidepressants).

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Pain ratings for heat stimuli | 3 years
  A 30-second tonic heat pain at the intensity of 46°C will be delivered to the volar forearm. During the heat stimulus, pain intensity ratings will be obtained.
Pain ratings for cold stimuli | 3 years
  Immersion of the foot into a cold water bath (8°C). Pain ratings of the water immersion will be collected at the end of the immersion.
Conditioned pain modulation | 3 years
  The CPM paradigm assesses endogenous inhibitory pain modulation efficiency related to spatial filtering of nociceptive information. CPM testing includes the application of a "test" stimulus without conditioning (control run) and a subsequent application of the same test stimulus together with a conditioning stimulus (conditioning run). The difference in pain sensitivity between the control and the conditioning run is the CPM response The test stimulus will be A 30-second tonic heat pain at the intensity of 46°C will be delivered to the volar forearm, and pressure pain thresholds at the trapezius.
  The conditioning stimulus will be immersion of the foot into a cold water bath (8°C). Pain ratings of the water immersion will be collected at the end of the immersion.
Testosterone levels | 3 years
  A blood draw will be collected, and total testosterone levels will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Nahman-Averbuch, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided